CLINICAL TRIAL: NCT05346133
Title: Adapting the Suicide Safety Planning Intervention for Delivery to Adolescents in Mozambican Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathryn L. Lovero, PhD, Assistant Professor of Sociomedical Sciences, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8129; K01MH120258 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Suicide; Adolescent Behavior
MeSH Terms: conditions — Suicide; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPI-A Adolescents (Other): Adolescents with moderate risk will receive the SPI-A intervention from the provider. Adolescents with high risk will be immediately taken to the mental health specialist at the primary care clinic. Following creation of the safety plan, patients are followed-up with at least twice to assess risk and review their plan. Following completion of the pilot, the investigators will interview all included providers as well as 18 adolescents who participated in SPI-A and their caregivers.
  Interventions: Behavioral: Suicide Prevention Intervention for Adolescents

INTERVENTIONS:
Behavioral: Suicide Prevention Intervention for Adolescents — Suicide Safety Planning Intervention (SPI). SPI is a very brief intervention (20-45 minutes) that provides patients with specific strategies to use to decrease the risk of suicidal behavior. SPI begins with psychoeducation about suicide risk, then the clinician and patient collaboratively create a stepwise plan that includes a simple list of individually tailored, concrete coping mechanisms to be enacted during or leading up to a crisis. The steps of the safety plan include: 1) recognizing warning signs of a crisis; 2) employing internal coping strategies; 3) using social contacts and settings to distract from suicidal thoughts; 4) seeking help from family members or close friends; 5) contacting healthcare or emergency services; and 6) reducing access to means. SPI providers work with caregivers to help them monitor warning signs of suicide risk, encourage the use of the safety plan by their adolescent, and reduce access to lethal means in the home.

SUMMARY:
Globally, suicide is ranked as the second leading cause of death for youth ages 10-24 years, and more than 75% of all deaths by suicide occur in low- and middle-income countries (LMIC). However, the vast majority of adolescents in LMIC do not have access to mental health care, and contextually appropriate strategies for delivering evidence-based interventions for managing suicide risk are needed to expand services to these areas. In the present study, the investigators will adapt and pilot test the Suicide Safety Planning Intervention for Adolescents (SPI-A) delivered by primary care providers in Mozambique, an LMIC in southeastern Africa.

DETAILED DESCRIPTION:
The investigators will provide a day-long training in SPI-A to 12 adolescent healthcare providers at 2 primary care clinics. Following the training, the providers will participate in a workshop with the research team to adapt SPI-A to their clinic setting, focusing on any SPI-A content modifications required for local adolescents (e.g. relevant examples of suicide risk warning signs), developing procedures for safe management of adolescents with imminent suicide risk in their clinic, strategies for engaging caregivers, and follow-up procedures. Providers will then be certified in SPI-A following 6-weeks of supervision.

After providers are certified in SPI-A, the intervention will be pilot tested in their primary care facilities. Providers will use a standardized questionnaire to screen included adolescents for suicide risk at the end of their clinic visit. Adolescents with moderate risk will receive the SPI-A intervention from the provider. Adolescents with high risk will be immediately taken to the mental health specialist (psychologist or psychiatrist) at the primary care clinic. Enrollment of participants will continue until each of the 12 primary care providers has completed SPI-A with 2 adolescents (n=24 adolescents completing SPI-A in total). Based on previous research exploring the prevalence of suicide risk in this adolescent population, the investigators anticipate needing to include 200 adolescents in total to be screened for suicide risk to identify 24 with moderate risk that will participate in SPI-A. Following completion of the pilot, the investigators will interview all included providers as well as 18 adolescents who participated in SPI-A and their caregivers. The goal of the trial is to determine 1) how primary care providers feel about delivering SPI-A, 2) how adolescents feel about participating in SPI-A, and 3) whether SPI-A results in reduced suicide risk levels in Mozambican adolescents.

ELIGIBILITY:
Adolescents:

Inclusion Criteria:

* Ages 12-19
* Portuguese-speaking
* Provide informed assent (ages 12-17) or consent (ages 18-19)
* Caregiver provides permission to participate (ages 12-17) Interview Interview

Exclusion Criteria:

* Having acute illness which requires immediate continued care
* Lacking lack of capacity/cognitive impairment for assent

Caretaker:

Inclusion Criteria:

* Parent or guardian of participating adolescent
* Present with adolescent at intervention clinics
* Portuguese-speaking
* Provide permission for adolescent participation Provide informed consent

Exclusion Criteria:

* Lacking lack of capacity/cognitive impairment for assent

Provider:

Inclusion Criteria:

- Providers in adolescent services at intervention clinics

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Change in suicide risk | 1 month
  Measuring change in suicide risk as measured by the "Columbia-Suicide Severity Rating Scale" (abbreviated as C-SSRS) at baseline (inclusion) and after 1 month.
  Scores range from 1-3 with 1 being low risk (the better outcome), 2 being moderate risk, and 3 being high risk (the worse outcome).

SECONDARY OUTCOMES:
Frequency of Suicide Safety Plan use | 1 month
  Frequency of Suicide Safety Plan use, measured by the question "In the past week, how often have you used your safety plan?" 1-month post inclusion. The outcomes range from 0-4, with 0 being "never" and 4 being "more than once a day."

OTHER OUTCOMES:
Frequency of use of specific coping behaviors. | 1 month
  Frequency of use of specific coping behaviors scores range from 0-2 with 2 being the better outcome (more use of coping behaviors). The average of scores is calculated across six of the following questions: "1. Try to tell yourself something calming or positive?", "2. Try to relax or do something calming?", "3. Think about reasons for living?", "4. Talk to a family member?", "5. Talk to a friend or another support person?", "6. Talk to a therapist, counselor, or doctor?", "7. Seek out emergency services?" with the answers options being never (0), sometimes (1), and always (2).

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lovero, PhD, Principal Investigator — Columbia University
Locations (2):
- Mozambique (2):
  - Centro de Saude Alto Mae, Maputo
  - Centro de Saude Bagamoio, Maputo

IPD SHARING:
Plan to Share IPD: No